CLINICAL TRIAL: NCT00988104
Title: Preventing Long Term Psychiatric Disability Among Those With Major Burn Injuries: the Safety, Meaning, Activation and Resilience Trial (SMART)
Brief Title: Preventing Long Term Psychiatric Disability Among Those With Major Burn Injuries
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA_00002545; NIDRR H133A070045; H133A070045 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Stress Disorders, Post-Traumatic; Mood Disorders; Sleep Disorders
Keywords: Behavior Therapy; Randomized Controlled Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mood Disorders; Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Supportive Counseling (Active Comparator)
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT (4 sessions): 1) Cognitive therapy targeting key appraisals. 2) Prolonged exposure targeting trauma memories and reminders. 3) Active coping/Anxiety Management training mindfulness-based techniques.
  Other Names: SMART
  Arms: Cognitive Behavioral Therapy
Behavioral: Supportive Counseling — Supportive counseling (4 sessions): common factors among effective psychotherapies (e.g., empathy, positive regard)
  Other Names: Usual Care
  Arms: Supportive Counseling

SUMMARY:
The purpose of this study is to determine whether a newly developed, brief cognitive behavioral intervention, relative to supportive counseling, is effective in reducing acute stress disorder (ASD) and preventing post traumatic stress disorder (PTSD) and depression.

DETAILED DESCRIPTION:
Importance: Burns are painful, life threatening and disfiguring. Severe psychological distress, pain and sleep disturbance are among the most common, enduring and disabling of secondary complications, however, no evidence based treatments exists for these complex problems in the acute burn care setting.

Design: Randomized, controlled effectiveness trial, group assignment blinded to baseline status, groups stratified by history of pre-existing psychiatric disorder.

Objectives. To develop the Safety, Meaning, Activation and Resilience Training (SMART) protocol; To evaluate its short and long-term effectiveness, relative to viable placebo, Supportive Counseling (SC), in improving key dependent measures (e.g., ASD, PTSD), mediators, and, enhancing health and function outcomes.

Setting: A leading edge, State-dedicated, regional burn center in a major, metropolitan teaching hospital serving diverse residents from large urban settings, small towns and remote rural areas.

Interventions: SMART (focused cognitive-behavioral therapy with training in anxiety management, and treatment with prolonged exposure and cognitive restructuring) will be contrasted with SC (non-directive empathy, warmth, positive regard).

Primary Outcome Measures: Health (psychological distress, sleep, pain), function (physical, psychological, social), costs (direct and indirect).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* acute burn injury
* exceeding criteria on screening instrument at baseline (in-hospital prior to treatment): Acute Stress Disorder Scale (ASDS score ≥ 37: acute posttrauma distress).

Exclusion Criteria:

* Age less than 18 or greater than 70 years
* Presence of a significant cognitive / neurological or psychiatric condition precluding informed consent (e.g., psychosis, acute suicidality)
* Inability to communicate in English
* intubated or sedated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10-16 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview for DSM IV: Mood and PTSD modules | 1 week, 1 month and 6 months post-treatment

SECONDARY OUTCOMES:
Davidson Trauma Scale | 1 week, 1 month and 6 months post-treatment
Patient Health Questionnaire - 9 (depression) | 1 week, 1 month and 6 months post-treatment
Insomnia Severity Index | 1 week, 1 month and 6 months post-treatment
Post Traumatic Growth Inventory | 1 week, 1 month and 6 months post-treatment
McGill pain Questionnaire | 1 week, 1 month and 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: James A Fauerbach, PhD, Principal Investigator — Johns Hopkins University; Una D McCann, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Burn Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] McKibben JB, Bresnick MG, Wiechman Askay SA, Fauerbach JA. Acute stress disorder and posttraumatic stress disorder: a prospective study of prevalence, course, and predictors in a sample with major burn injuries. J Burn Care Res. 2008 Jan-Feb;29(1):22-35. doi: 10.1097/BCR.0b013e31815f59c4. PMID 18182894
- [Background] Fauerbach JA, McKibben J, Bienvenu OJ, Magyar-Russell G, Smith MT, Holavanahalli R, Patterson DR, Wiechman SA, Blakeney P, Lezotte D. Psychological distress after major burn injury. Psychosom Med. 2007 Jun;69(5):473-82. doi: 10.1097/psy.0b013e31806bf393. PMID 17585064
- [Background] Smith MT, Klick B, Kozachik S, Edwards RE, Holavanahalli R, Wiechman S, Blakeney P, Lezotte D, Fauerbach JA. Sleep onset insomnia symptoms during hospitalization for major burn injury predict chronic pain. Pain. 2008 Sep 15;138(3):497-506. doi: 10.1016/j.pain.2008.01.028. Epub 2008 Mar 24. PMID 18362052
- [Background] Edwards RR, Magyar-Russell G, Thombs B, Smith MT, Holavanahalli RK, Patterson DR, Blakeney P, Lezotte DC, Haythornthwaite JA, Fauerbach JA. Acute pain at discharge from hospitalization is a prospective predictor of long-term suicidal ideation after burn injury. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S36-42. doi: 10.1016/j.apmr.2007.05.031. PMID 18036980
- [Background] Edwards RR, Smith MT, Klick B, Magyar-Russell G, Haythornthwaite JA, Holavanahalli R, Patterson DR, Blakeney P, Lezotte D, McKibben J, Fauerbach JA. Symptoms of depression and anxiety as unique predictors of pain-related outcomes following burn injury. Ann Behav Med. 2007 Nov-Dec;34(3):313-22. doi: 10.1007/BF02874556. PMID 18020941
- [Background] Esselman PC, Thombs BD, Magyar-Russell G, Fauerbach JA. Burn rehabilitation: state of the science. Am J Phys Med Rehabil. 2006 Apr;85(4):383-413. doi: 10.1097/01.phm.0000202095.51037.a3. No abstract available. PMID 16554686
- [Background] Fauerbach JA, Lezotte D, Hills RA, Cromes GF, Kowalske K, de Lateur BJ, Goodwin CW, Blakeney P, Herndon DN, Wiechman SA, Engrav LH, Patterson DR. Burden of burn: a norm-based inquiry into the influence of burn size and distress on recovery of physical and psychosocial function. J Burn Care Rehabil. 2005 Jan-Feb;26(1):21-32. doi: 10.1097/01.bcr.0000150216.87940.ac. PMID 15640730
- [Background] Lawrence JW, Fauerbach JA. Personality, coping, chronic stress, social support and PTSD symptoms among adult burn survivors: a path analysis. J Burn Care Rehabil. 2003 Jan-Feb;24(1):63-72; discussion 62. doi: 10.1097/00004630-200301000-00016. PMID 12543997
- [Background] Fauerbach JA, Richter L, Lawrence JW. Regulating acute posttrauma distress. J Burn Care Rehabil. 2002 Jul-Aug;23(4):249-57. doi: 10.1097/00004630-200207000-00005. PMID 12142577
- [Background] Fauerbach JA, Lawrence JW, Fogel J, Richter L, Magyar-Russell G, McKibben JB, McCann U. Approach-avoidance coping conflict in a sample of burn patients at risk for posttraumatic stress disorder. Depress Anxiety. 2009;26(9):838-50. doi: 10.1002/da.20439. PMID 19170120
- See also: Johns Hopkins Burn Center — http://www.hopkinsmedicine.org/burn/index.html